CLINICAL TRIAL: NCT05765201
Title: Phacoemulsification at High IOP and Physiologic IOP: Impact on Anterior and Posterior Segment Physiology
Status: Completed | Type: Observational
Sponsor: Matthew Rauen (Other)
Responsible Party: Sponsor-Investigator, Matthew Rauen, MD, Wolfe Eye Clinic
Organization: Wolfe Eye Clinic (Other)
Other Study IDs: Alcon IIT # 75098433
Record Dates: First submitted 2023-01-17; First posted 2023-03-13 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Nuclear Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High IOP: Eyes in this arm will maintain an IOP of 65mmHg throughout the cataract surgery.
  Interventions: Other: High IOP
- Low IOP: Eyes in this arm will maintain an IOP of 28mmHg throughout the cataract surgery.
  Interventions: Other: Low IOP

INTERVENTIONS:
Other: High IOP — Prospective, single-surgeon, randomized, paired-eye study; patients undergoing sequential, uncomplicated bilateral phacoemulsification using Active Sentry handpiece® with intraocular IOP ≤ 28mmHg (low IOP) in one eye and with IOP ≥ 60mmHg (high IOP) in the other eye
  Groups: High IOP
Other: Low IOP — Prospective, single-surgeon, randomized, paired-eye study; patients undergoing sequential, uncomplicated bilateral phacoemulsification using Active Sentry handpiece® with intraocular IOP ≤ 28mmHg (low IOP) in one eye and with IOP ≥ 60mmHg (high IOP) in the other eye
  Groups: Low IOP

SUMMARY:
The purpose of this study is to investigate the anterior and posterior structure and functional changes and vascular alterations when performing phacoemulsification at high IOP vs low, more physiological IOP using Centurion® Vision System with Active Sentry® handpiece. These devices are approved by the US Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
To investigate the anterior and posterior physiological changes when performing phacoemulsification at high IOP vs low, more physiologic IOP using Centurion® Vision System with Active Sentry® handpiece

Prospective, single-surgeon, randomized, paired-eye study; patients undergoing sequential, uncomplicated bilateral phacoemulsification using Active Sentry handpiece® with intraocular IOP ≤ 28mmHg (low IOP) in one eye and with IOP ≥ 60mmHg (high IOP) in the other eye

Operating at lower, more physiological IOP using Active Sentry® handpiece during cataract surgery will use less BSS fluid usage. (Lower IOP settings are also expected to result in less subclinical changes).

ELIGIBILITY:
Inclusion Criteria:

* No prior ocular surgery including corneal refractive surgery
* Bilateral visually significant cataract, similar in density (LOCS III grade 2+), undergoing uncomplicated cataract surgery
* Equal dilated pupil size ≥6mm, no use of pupil expansion devices
* Unremarkable systemic health but inclusive of controlled type II diabetes and hypertension with normal OCT angiography at baseline
* A1C ≤ 8% on single monotherapy or lifestyle adjustments
* To maintain high sensitivity/specificity, patients to fall under OCT normative database:
* Axial length 22-26mm
* Refractive error between -5.00D to +5.00D
* Cylinder ≤ 3.00D
* Normal K values <47.00D
* Axial eye length cannot vary by more than 0.4 mm in an individual patient
* Normal CCT range 540µm ± 50

Exclusion Criteria:

* H/o corneal disease or dystrophies
* Media opacification for reasons other than cataract
* Compromised zonular integrity or stability
* Retinal and retinal vascular pathologies, age-related macular degeneration
* Glaucoma
* Patients with uncontrolled systematic diseases; including hypertension, diabetes, systemic cardiovascular diseases and hematological diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 25 cataract surgery patients form ophthalmology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Estimated fluid usage- High IOP Group | Intraoperative
  Measurement of fluid usage (ml).
Estimated fluid usage- Low IOP Group | Intraoperative
  Measurement of fluid usage (ml).

SECONDARY OUTCOMES:
Macular Thickness | post procedure at 1 week, 1 month, and 3 months
  Macular thickness measured in microns at week 1, month 1, and month 3. Measured by optical coherence tomography (OCT).
Corneal Thickness | post procedure at 1 day, 1 week, 1 month, and 3 months
  Corneal thickness measured in microns at 1 day, week 1, month 1, and month 3. Measured by pentacam tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rauen, MD, Principal Investigator — Wolfe Eye Clinic
Locations (1):
- Wolfe Eye Clinic, West Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tang Y, Chen X, Zhang X, Tang Q, Liu S, Yao K. Clinical evaluation of corneal changes after phacoemulsification in diabetic and non-diabetic cataract patients, a systematic review and meta-analysis. Sci Rep. 2017 Oct 26;7(1):14128. doi: 10.1038/s41598-017-14656-7. PMID 29074989
- [Result] Li T, Guadie A, Feng L, Fan J, Jiang Z, Liu F. Influence of cataract surgery on macular vascular density in patients with myopia using optical coherence tomography angiography. Exp Ther Med. 2020 Dec;20(6):258. doi: 10.3892/etm.2020.9388. Epub 2020 Oct 27. PMID 33199984
- [Result] Zeng S, Liang C, He Y, Chen Y, Zhao Q, Dai S, Cheng F, Zhang J, Jiang X. Changes of Subfoveal Choroidal Thickness after Cataract Surgery: A Meta-Analysis. J Ophthalmol. 2018 Nov 12;2018:2501325. doi: 10.1155/2018/2501325. eCollection 2018. PMID 30607294
- [Result] Vasavada V, Raj SM, Praveen MR, Vasavada AR, Henderson BA, Asnani PK. Real-time dynamic intraocular pressure fluctuations during microcoaxial phacoemulsification using different aspiration flow rates and their impact on early postoperative outcomes: a randomized clinical trial. J Refract Surg. 2014 Aug;30(8):534-40. doi: 10.3928/1081597X-20140711-06. PMID 25325894
- [Result] Chen D, Zhu J, Li J, Ding XX, Lu F, Zhao YE. Effect of simulated dynamic intraocular pressure on retinal thickness measured by optical coherence tomography after cataract surgery. Int J Ophthalmol. 2012;5(6):687-93. doi: 10.3980/j.issn.2222-3959.2012.06.07. Epub 2012 Dec 18. PMID 23275902
- [Result] Liu X, Fang Y, Zhou Y, Wang M, Luo Y. Dynamic changes in retinal vessel density observed by optical coherence tomography angiography after phacoemulsification: active vs gravity fluidics system. Arq Bras Oftalmol. 2022 Apr 8;85(2):205-207. doi: 10.5935/0004-2749.20220093. eCollection 2022. No abstract available. PMID 35416902